CLINICAL TRIAL: NCT02341157
Title: Implementation, Compliance, and Effectiveness of Integrating the PikoLogic® Into Disease Management Discharge Care for Patients With COPD Exacerbation: A Prospective Cohort Study.
Brief Title: ICE COPD PikoLogic® Cohort Study.Implementation, Compliance, and Effectiveness of Integrating the PikoLogic®
Acronym: ICE
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left the University of Louisville.
Sponsor: University of Louisville (Other)
Collaborators: nSpire Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NSH 002-00
Record Dates: First submitted 2014-12-18; First posted 2015-01-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2015-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a two-step observational cohort study evaluating the impact of adding PikoLogic® to the current disease management COPD discharge protocol subsequent to an admission for COPD exacerbation.

DETAILED DESCRIPTION:
Candidate subjects participating in the cohort study will receive training by the clinical research associate (CRA) on the use of PikoLogic® for home disease management prior to discharge from the hospital. The CRA will also confirm COPD discharge education was completed by a discharge coordinator and the patient understood the instructions. The CRA will review "seek medical care if:" and "seek immediate medical care if:" instructions at discharge. The discharge CRA will also evaluate subjects for their ability to use the PikoLogic® correctly and will score the patient using an objective and subjective measurement tool. A modified Discharge Knowledge Assessment Tool© will be utilized.1 Objective measurements will include training time and patient compliance with PikoLogic® prior to discharge. Subjective data scores and objective measurements will be utilized for program implementation evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of COPD at or prior to hospitalization.
2. Be hospitalized for one of the following reasons:

   * COPD exacerbation
   * COPD
   * COPD with pneumonia
3. Be an ex-smoker or current smoker with a smoking history of ≥ 10 pack years (i.e., 1 pack [20 cigarettes] per day for 10 years).
4. Be judged by the investigator to be in stable health (except for COPD variability) on the basis of medical history, physical examination, and routine laboratory data, and appears able to successfully complete this study.
5. Be willing to perform daily objective and subjective measurements using the PikoLogic® device and maintain daily utilization for 1 year following discharge.
6. The subject is fluent in English for reading and writing.
7. The subject provides written informed consent for the trial.

Exclusion Criteria:

1. Has a current diagnosis of any disease with chronic airflow obstruction other than COPD.
2. Is unwilling to use the PikoLogic® and unwilling to maintain a written record of hospitalization for 1 year.
3. Lives in a neighborhood with poor or no cellular coverage.
4. Is currently homeless or in jeopardy of being homeless during the 1 year study period.
5. Does not have a means to be transported to the follow up study visits.
6. Cannot be contacted easily.
7. Discharges against medical advice.
8. In hospice within one year prior to admission.
9. Is associated with the administration of the study. No family member of the investigational study staff may participate in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Have a diagnosis of COPD at or prior to hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
: patient diary compliance at 30 and 365 days post-discharge. | 30 days and 365 day reviews
  To evaluate short term clinical implementation and patient compliance of a COPD PikoLogic® discharge action plan for COPD patients to assist in home care self-monitoring.

SECONDARY OUTCOMES:
Time to first severe exacerbation, as defined by an event requiring hospitalization or evaluation in the emergency department 30 days to 1 year after enrollment. | 30 Days
Number of severe exacerbations, as defined by an event requiring hospitalization or evaluation in the emergency department 30 days to 1 year after enrollment. | 30 and 365 Days
Cost of care, defined as patient healthcare resource utilization and hospital charges if readmission occurs, in the 1 year (52 weeks) following 30 days from hospital discharge for treatment of COPD exacerbation. | 30 and 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Rodney J Folz, MD, PhD, Study Director — University of Louisville; Hiram Rivas-Perez, MD, Principal Investigator — University of Louisville